CLINICAL TRIAL: NCT06945016
Title: MOnitoring NUtritional COnsequences of Obesity Treatment on Women's Health and Transgenerational Effects for Healthier Future Generations: a Multicentre Prospective Observational Cohort Study
Brief Title: Monitoring Nutritional Consequences of Obesity Treatment on Women's Health
Acronym: MONUCO
Status: Recruiting | Type: Observational
Sponsor: Wageningen University and Research (Other)
Collaborators: Rijnstate Hospital (Other)
Responsible Party: Principal Investigator, Agnes Berendsen, Assistant Professor, Wageningen University and Research
Other Study IDs: NL86647.091.24
Record Dates: First submitted 2025-02-12; First posted 2025-04-25 (Actual); Last update posted 2025-07-10 (Actual); Status verified 2025-04

CONDITIONS: Obesity and Obesity-related Medical Conditions; Bariatric Surgery; Anti-obesity Agents; Body Composition; Muscle Strength; Reproductive Health; Mental Health; Pregnancy; Nutritional Status
Keywords: cohort; obesity treatment; obesity; Bariatric surgery; anti-obesity agents; body composition; nutrition; observational
MeSH Terms: conditions — Obesity; Psychological Well-Being

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — The following samples will be retained: urine, stool, venous blood (serum, plasma and full blood), cord blood and breastmilk.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- General cohort: Women aged 18-55 years of age living with obesity (BMI => 30kg/m2) undergoing either surgical (RYGB, OAGB, SG) or pharmacological obesity treatment.
- Birth cohort: Pregnant women aged 18-45 years of age having received prior obesity treatment, either surgical (RYGB, OAGB, SG) or pharmacological for at least 4 months under medical supervision (any type)

SUMMARY:
The goal of this observational study is to investigate the long-term effect of obesity treatments on the health of women. This study will specifically focusses on the effects on nutritional intake, nutritional status, musculoskeletal health and reproductive health. Additionally, this study will also investigate the effect of obesity treatment on pregnancy outcomes and child development.

To achieve the goal of this study, participants already receiving either surgical treatment for obesity or treatment with anti-obesity medication as part of their regular medical care will fill in additional questionnaires, provide blood, urine and feces samples, and undergo additional measurements of body composition and muscle strength up to for 10 years.

DETAILED DESCRIPTION:
The MONUCO study is a multicenter 10-year prospective observational cohort study with an integrated birth cohort. Women between the ages of 18-55 years approved for either surgical or pharmacological obesity treatment at one of the participating centers are invited. Follow-up data will be collected at 6-weeks pre-treatment, three months, six months and one year up to ten years post-surgery. At each time point, participants fill in questionnaires on lifestyle factors, gastrointestinal complaints, menstrual and postmenopausal complaints, and mental health. They also record their dietary intake using FFQ's and a 2h-recall method via the Traqq application. Additionally, they provide blood, urine and feces samples which are stored at -80 degrees Celsius for future analysis. During a study visit at each time point, height, weight, hip and waist circumference is measured as well as body composition with BIA and muscle strength and balance with handgrip strength and a timed chair-stand test. In a subgroup of the study population, a DEXA scan and/or MRI scan is performed and physical activity is tracked with an accelerometer.

Women who become pregnant during the follow-up period will be included in the integrated birth cohort. To supplement this number, pregnant women who have had obesity treatment who are not a part of the overall cohort are also invited. Within the integrated birth cohort, measurements are collected at each trimester during pregnancy and two months post-partum, six months post-partum, after one year up to four years after pregnancy. During pregnancy, the participant fill in questionnaire on lifestyle factors, gastrointestinal complaints and pregnancy-related complaints as well as record dietary intake with an FFQ and 2h-recall method. In this group also provides blood, urine, stool and human milk samples.

ELIGIBILITY:
General Inclusion Criteria:

* Female sex at birth
* Aged 18-55 years of age
* Living with obesity (BMI ≥ 30 kg/m2)
* Approved for obesity treatment in one of the participating hospitals:
* Undergoing primary bariatric surgery (RYGB, OAGB or SG)
* Receiving obesity medication (any type) with a BMI ≥30 kg/m2 under medical supervision.
* For those undergoing MRI, DEXA and quantitative ultrasound scan: Willing to be informed about incidental findings of pathology and approving of reporting this to their general physician.

Additional inclusion criteria for birth cohort:

* Being pregnant
* Age 18-45 years of age
* Having received prior obesity treatment, either surgical (RYGB, OAGB, SG) or pharmacological for at least 4 months under medical supervision (any type).

General Exclusion Criteria:

* Male sex at birth
* Aged <18 or >55 years of age
* BMI <30 kg/m2
* Not able to read and/or write in Dutch
* Undergoing a revisional or secondary bariatric procedure (excluding previous gastric banding)
* Malnutrition due to other chronic condition, specifically malignancy, substance abuse
* (mental) condition that makes it impossible to fill out a questionnaire correctly.
* For those undergoing a DEXA scan: height >196 cm or weight >160 kg
* For those undergoing a MRI scan: having a contra-indication to MRI scanning including (but not limited to) pacemakers and defibrillators, intraorbital or intraocular metallic fragments, ferromagnetic implans or claustrophobia.

Additional exclusion criteria birth cohort:

* Aged <18 or >45 years of age
* >25 weeks of gestation
* Multiple pregnancy
* Reversal of the bariatric procedure

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: The study population of the MONUCO study consists of women undergoing either surgical or pharmacological obesity treatment. Participants who become pregnant during the general cohort will be asked to participate within the birth cohort. Additionally, all other women with a history of obesity treatment and who are pregnant are eligible to participate in the birth cohort as well.
  Patient recruitment will start at Vitalys, a clinic for obesity treatment, part of Rijnstate hospital, with locations in Arnhem/Elst and Ede (Ziekenhuis Gelderse Vallei). Recruitment will be expanded to other high-volume obesity centres in the Netherlands.
Sampling Method: Non-Probability Sample
Enrollment: 1150 (Estimated)
Dates: Start 2025-01-28 (Actual); Primary Completion 2040-01-28 (Estimated); Study Completion 2040-01-28 (Estimated)

PRIMARY OUTCOMES:
Body composition analysis | Assessed at baseline, and at 3 months, 6 months 1 year, 2 years, 3 years, 4 years, 5 years and 10 years post surgery or pharmacological treatment initiation. In the birth cohort it is additionally assessed at 1 year post-partum.
  The analysis of body composition parameters using bioelectrical impedance analysis (BIA). Raw BIA parameters such as reactance, resistance and phase angle as well as derived parameters including fat-free mass, fat mass and total body water are recorded.
Handgrip strength | Assessed at baseline, and at 3 months, 6 months 1 year, 2 years, 3 years, 4 years, 5 years and 10 years post surgery or pharmacological treatment initiation. In the birth cohort it is additionally assessed at 1 year post-partum.
  Maximal handgrip strength out of three repetitions with both the dominant and non-dominant hand.
Timed Chair-stand-test/Five Times Sit to Stand test | Assessed at baseline, and at 3 months, 6 months 1 year, 2 years, 3 years, 4 years, 5 years and 10 years post surgery or pharmacological treatment initiation. In the birth cohort it is additionally assessed at 1 year post-partum.
  The time in seconds it takes a participant to stand-up from a seated position and sit-down 5 times without using their hands.
Bone mineral density | Assessed at baseline, and at 6 months, 1 year, 2 years, 3 years, 4 years, 5 years, and 10 years post surgery or pharmacological treatment initiation.
  Total body and hip bone mineral density measured with a DEXA scan.
Lean mass | Assessed at baseline, and at 6 months, 1 year, 2 years, 3 years, 4 years, 5 years, and 10 years post surgery or pharmacological treatment initiation.
  Total lean mass and appendicular lean mass assessed with a DEXA scan.
Peak torque of knee extensors and flexors | Assessed at baseline, and at 6 months, 1 year, 2 years, 3 years, 4 years, 5 years, and 10 years post surgery or pharmacological treatment initiation.
  The maximum of 5 repetitions at a constant angle speeds of 60 degrees per second in an isokinetic dynamometer.
Total work of knee extensors and flexors | Assessed at baseline, and at 6 months, 1 year, 2 years, 3 years, 4 years, 5 years, and 10 years post surgery or pharmacological treatment initiation.
  The work accomplished during 15 repetitions at 180 degrees/second in a isokinetic dynamometer.
Bone formation | Assessed at baseline, and at 6 months, 1 year, 2 years, 3 years, 4 years, 5 years, and 10 years post surgery or pharmacological treatment initiation. In the birth cohort additionally during first and third trimester and at 1 year post-partum.
  P1NP (Total procollagen type 1-teriminal propeptide) measured in a venous blood sample.
Bone resorption | Assessed at baseline, and at 6 months, 1 year, 2 years, 3 years, 4 years, 5 years, and 10 years post surgery or pharmacological treatment initiation. In the birth cohort additionally during first and third trimester and at 1 year post-partum.
  CTX (type-1 collagen) measured in a venous blood sample.
Proton density fraction in the bone marrow | Assessed at baseline, and at 6 months, 2 years, 4 years post surgery or pharmacological treatment initiation.
  The proton density fat fraction of the bone marrow obtained through an MRI scan.
Proton density fraction in the muscles of the thigh and back | Assessed at baseline, and at 6 months, 2 years, 4 years post surgery or pharmacological treatment initiation.
  The proton density fat fraction of the muscle in the low back and upper thigh obtained through an MRI scan.
Habitual dietary intake | Assessed at baseline, and 1 year, 2 years, 3 years, 4 years, 5 years and 10 years post surgery or pharmacological treatment initiation.
  Assessed through a food-frequency questionnaire.
Actual dietary intake | At 3 months and 6 months post surgery or pharmacological treatment initiation. In the birth cohort additionally during first and third trimester and at 2 months post-partum.
  Assessed with the TRAQQ app, a mobile phone application that performs 9 2 -h recalls on 3 days.
Nutrient status | Assessed at baseline, and at 6 months, 1 year, 2 years, 3 years, 4 years, 5 years, and 10 years post surgery or pharmacological treatment initiation. In the birth cohort during first, second and third trimester and at 2 months and 1 year post-partum.
  Presence of nutrient deficiencies.
Neonatal birth weight | Directly after birth
  Neonatal birth weight, weight-for-age percentile and classification of small-for-gestational age.
Calcaneal Speed of Sound | Assessed during first trimester, third trimester and 1 year post-partum.
  Speed of Sound in measured in the calcaneus with a quantitative ultrasound machine.
Calcaneal Broadband Ultrasound Attenuation | Assessed during first trimester, third trimester and 1 year post-partum.
  Broadband ultrasound attenuation in measured in the calcaneus with a quantitative ultrasound machine.
Diet quality | Assessed in the birth cohort during the second trimester and at 1 years and 4 years post-partum.
  Assessed through the Eetscore, a brief food-frequency questionnaire.
Neonatal nutrient status | Assessed in the birth cohort at birth.
  Presence of nutrient deficiencies measured in cord blood collected after birth.
Fetal growth: biparietal diameter | Assessed in first trimester, second trimester and third trimester.
  Biparietal diameter measured during prenatal ultrasounds.
Fetal growth: abdominal circumference | Assessed in first trimester, second trimester and third trimester.
  Abdominal circumference measured during the prenatal ultrasounds.
Fetal growth: femur length | Assessed in first trimester, second trimester and third trimester.
  Femur length measured during the prenatal ultrasounds.
Fetal growth: head circumference | Assessed in first trimester, second trimester and third trimester.
  Head circumference measured during the prenatal ultrasounds.
Fetal growth: frontal occipital diameter | Assessed in first trimester, second trimester and third trimester.
  Frontal occipital diameter measured during the prenatal ultrasounds.
Estimated fetal weight | Assessed in first trimester, second trimester and third trimester.
  Estimated based on prenatal ultrasounds.

SECONDARY OUTCOMES:
General information on child growth and development | Assessed at 2 months, 1 year and 4 years post-partum.
  Participants in the birth cohort will fill in a general questionnaire with questions about body length, height and weight as well as other developmental aspects.
Sleep quality | Assessed at baseline, and at 6 months, 1 year, 2 years, 3 years, 4 years, 5 years, and 10 years post surgery or pharmacological treatment initiation. In the birth cohort it is assessed during second trimester and at 1 year post-partum.
  Assessed using the Pitsburg Sleep Quality Index (PSQI). The minimum and maximum values of this index are 0 and 21 respectively. Higher scores indicate poorer sleep quality.
Physical activity | Assessed at baseline, and at 6 months, 1 year, 2 years, 3 years, 4 years, 5 years, and 10 years post surgery or pharmacological treatment initiation. In the birth cohort it is assessed during second trimester and at 1 year post-partum.
  Assessed using the Short QUestionnaire to ASsess Health-enhancing physical activity (SQUASH). The results can be expressed as minutes per week spend on physical activity or a metabolic equivalent task (MET) score. A higher MET score indicates more intense physical activity. The minimum MET score is 1. There is no official upper limit of the MET score.
Sleep time | Assessed at baseline, and at 6 months, 1 year, 2 years, 3 years, 4 years, 5 years, and 10 years post surgery or pharmacological treatment initiation.
  Assess using an accelerometer (Actigraph). The accelerometer was worn during 7 days at each follow-up measurement.
Energy expenditure (kcals) | Assessed at baseline, and at 6 months, 1 year, 2 years, 3 years, 4 years, 5 years, and 10 years post surgery or pharmacological treatment initiation.
  Assess using an accelerometer (Actigraph). The accelerometer was worn during 7 days at each follow-up measurement.
Steps | Assessed at baseline, and at 6 months, 1 year, 2 years, 3 years, 4 years, 5 years, and 10 years post surgery or pharmacological treatment initiation.
  Assess using an accelerometer (Actigraph). The accelerometer was worn during 7 days at each follow-up measurement.
Metabolic Equivalent of Task (MET) rate | Assessed at baseline, and at 6 months, 1 year, 2 years, 3 years, 4 years, 5 years, and 10 years post surgery or pharmacological treatment initiation.
  Assess using an accelerometer (Actigraph). The accelerometer was worn during 7 days at each follow-up measurement.
Total sedentary time | Assessed at baseline, and at 6 months, 1 year, 2 years, 3 years, 4 years, 5 years, and 10 years post surgery or pharmacological treatment initiation.
  Assess using an accelerometer (Actigraph). The accelerometer was worn during 7 days at each follow-up measurement.
Total time doing light physical activity | Assessed at baseline, and at 6 months, 1 year, 2 years, 3 years, 4 years, 5 years, and 10 years post surgery or pharmacological treatment initiation.
  Assess using an accelerometer (Actigraph). The accelerometer was worn during 7 days at each follow-up measurement.
Total time doing moderate physical activity | Assessed at baseline, and at 6 months, 1 year, 2 years, 3 years, 4 years, 5 years, and 10 years post surgery or pharmacological treatment initiation.
  Assess using an accelerometer (Actigraph). The accelerometer was worn during 7 days at each follow-up measurement.
Total time doing vigorous physical activity | Assessed at baseline, and at 6 months, 1 year, 2 years, 3 years, 4 years, 5 years, and 10 years post surgery or pharmacological treatment initiation.
  Assess using an accelerometer (Actigraph). The accelerometer was worn during 7 days at each follow-up measurement.
Menstrual complaints | Assessed at baseline, and at 6 months, 1 year, 2 years, 3 years, 4 years, 5 years, and 10 years post surgery or pharmacological treatment initiation. In the birth cohort it is assessed at 1 year post-partum.
  Assessed using a custom made questionnaire containing questions about menstrual history, dysmenorrhoea, menstrual complaints, bleeding and choice of contraceptives.
Menopausal complaints | Assessed at baseline, and at 6 months, 1 year, 2 years, 3 years, 4 years, 5 years, and 10 years post surgery or pharmacological treatment initiation. In the birth cohort it is assessed at 1 year post-partum.
  Assessed using a custom made questionnaire containing questions menopausal complaints and the use of hormones.
Gastrointestinal complaints | Assessed at baseline, and at 3 months, 6 months 1 year, 2 years, 3 years, 4 years, 5 years and 10 years post surgery or pharmacological treatment initiation. In the birth cohort it is assessed during the second trimester.
  Assessed with the gastrointestinal symptom rating scale (GSRS). The minimum score is 15 and the maximum score is 105. Higher score indicate worse gastrointestinal symptoms.
Irritable bowel syndrome related complaints | Assessed at baseline, and at 3 months, 6 months 1 year, 2 years, 3 years, 4 years, 5 years and 10 years post surgery or pharmacological treatment initiation. In the birth cohort it is assessed during the second trimester.
  Assessed with the Rome VI criteria.
Early dumping syndrome complaints | Assessed at 3 months, 6 months and 1 year post surgery or pharmacological treatment initiation. In the birth cohort it is assessed during the first and third trimester.
  Assessed with the Sigstad score. The mimimum and maximum values of the score are -5 and 25 respectively. Scores greater or equal to 7 indicate that dumping syndrome is likely. Higher scores indicates more and more severe dumping syndrome symptoms.
Dumping syndrome complaints | Assessed at 3 months, 6 months and 1 year post surgery or pharmacological treatment initiation. In the birth cohort it is assessed during the first and third trimester.
  Assessed with the Arts dumping score questionnaire. The minimum and maximum score of the score are 0 and 26 respectively. Higher scores indicate more severe dumping syndrome symptoms.
Food intolerances | Assessed at 3 months, 6 months and 1 year post surgery or pharmacological treatment initiation.
  Assessed with the quality of alimentation questionnaire.
Stool pattern | Assessed at baseline, and at 3 months, 6 months 1 year, 2 years, 3 years, 4 years, 5 years and 10 years post surgery or pharmacological treatment initiation. In the birth cohort it is assessed during the second trimester.
  Assessed with the Bristol stool chart. The chart indicates the form and consistency of the stool with 7 distinct types. From hard lumps (type 1) to watery stools (type 7).
Pregnancy related symptomes | Assessed in the birth cohort during first, second and third trimester.
  Assessed with the pregnancy symptoms inventory (PSI). This inventory include two subscales. The Frequency of Pregnancy Symptoms score ranges from 0 to 126, and the Limitation of Daily Activities score ranges from 42 to 126. Higher scores indicate more frequent symptoms and more severe limitation of daily activities.

OTHER OUTCOMES:
Obesity related quality of life | Assessed at baseline, and at 3 months, 6 months 1 year, 2 years, 3 years, 4 years, 5 years and 10 years post surgery or pharmacological treatment initiation.
  Assessed with a disease specific quality of life questionnaire called the OBESI-Q. The score ranges from 0 to 100 with higher scores indicating better quality of life.
Depression symptoms | Assessed at baseline, and at 3 months, 6 months 1 year, 2 years, 3 years, 4 years, 5 years and 10 years post surgery or pharmacological treatment initiation.
  Assessed with the Centre of Epidemiological Studies Depression Scale (CES-D). The score ranges from 0 to 60 with higher scores indicating more severe depressive symptoms.
Self-esteem | Assessed at baseline, and at 3 months, 6 months 1 year, 2 years, 3 years, 4 years, 5 years and 10 years post surgery or pharmacological treatment initiation.
  Assessed with the Rosenberg self-esteem scale (RSE). The score ranges between 0 and 30 with higher scores indicating better self-esteem.
Eating disorder symptoms | Assessed at baseline, and at 3 months, 6 months 1 year and 2 years post surgery or pharmacological treatment initiation. The score ranges from 0 to 6 with higher scores indicating more severe symptoms.
  Assessed with the eating disorder examination questionnaire (EDE-Q).
Post-partum depression risk | Assessed in the birth cohort at 2 months post-partum.
  Assessed with the Edinburg postnatal depression scale (EPDS). The score ranges from 0 to 30 with higher scores indicating more severe depression symptoms.
Gut microbiome composition | Assessed at baseline, and at 3 months, 6 months 1 year, 2 years, 3 years, and 5 years post surgery or pharmacological treatment initiation. In the birth cohort additionally at birth an 2 months post-partum in both mother and child.
  Assessed in by extracting DNA from collected stool samples.
Nutritional composition of human milk | Assessed at 2 months post-partum in the birth cohort.
  The macro and micronutrient content of human milk samples.
Urinary serotonine | Assessed at baseline, and at 6 months, 1 year, 2 years, 3 years, and 5 years post surgery or pharmacological treatment initiation. In the birth cohort additionally during first and second trimester and 2 months post-partum.
  Assessed in spot urine samples. The second urine of the day is collected.
Height | Assessed at baseline, and at 3 months, 6 months 1 year, 2 years, 3 years, 4 years, 5 years and 10 years post surgery or pharmacological treatment initiation. Additionally in the birth cohort during first, second, and third trimester.
  Height measured in cm with a stadiometer.
Waist circumference | Assessed at baseline, and at 3 months, 6 months 1 year, 2 years, 3 years, 4 years, 5 years and 10 years post surgery or pharmacological treatment initiation.
  Measured in cm at the midpoint between the top of the hip bone and bottom of the rib cage with a non-elastic tape measure. Average of two measurements is used.
Hip circumference | Assessed at baseline, and at 3 months, 6 months 1 year, 2 years, 3 years, 4 years, 5 years and 10 years post surgery or pharmacological treatment initiation.
  Measured in cm at the height of the greater trochanter with a non-elastic tape measure. Average of two measurements is used.
Weight | Assessed at baseline, and at 3 months, 6 months 1 year, 2 years, 3 years, 4 years, 5 years and 10 years post surgery or pharmacological treatment initiation. Additionally in the birth cohort during first, second, and third trimester.
  Weight measured in kg with calibrated scales.
General information | Assessed at baseline, and at 3 months, 6 months 1 year, 2 years, 3 years, 4 years, 5 years and 10 years post surgery or pharmacological treatment initiation.
  Participants complete a general questionnaire to gather information on sociodemographic factors, medical conditions or complications, medications, smoking, alcohol consumption and drug use.
General information pregnancy | Assessed during first, second and third trimester.
  Participants in the birth cohort complete a general questionnaire to gather information on sociodemographic factors, medical history, medications, smoking, alcohol consumption, drug use, and progression of the pregnancy.
Fat mass | Assessed at baseline, and at 6 months, 1 year, 2 years, 3 years, 4 years, 5 years, and 10 years post surgery or pharmacological treatment initiation.
  Total fat mass assessed with a DEXA scan.
Proton density fraction in the liver | Assessed at baseline, and at 6 months, 2 years, 4 years post surgery or pharmacological treatment initiation.
  The proton density fat fraction of the muscle in the liver obtained through an MRI scan.

CONTACTS AND LOCATIONS:
Overall Officials: Agnes Berendsen, PhD, Principal Investigator — Wageningen University and Research
Locations (1):
- Rijnstate Elst, Vitalys, Elst, Gelderland, Netherlands

IPD SHARING:
Plan to Share IPD: No
In due time, we plan to share all IPD that underlie results in a publication. However, as we have just started recruitment, no specific plans have been made yet. Once this is clear, we will update this registration.